CLINICAL TRIAL: NCT06274151
Title: Optimal Treatment of Inflammation Following Acute Skeletal Muscle Injury
Brief Title: Optimal Treatment of Acute Skeletal Muscle Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Monika Lucia Bayer, Senior Researcher, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-22038917
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Muscle Strain, Multiple Sites; Inflammation
MeSH Terms: conditions — Sprains and Strains; Inflammation | interventions — Naproxen; Anti-Inflammatory Agents, Non-Steroidal; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory medicine (Experimental): Week 2 after muscle strain injury Naproxen 500mg 2x daily
  Interventions: Drug: Naproxen 500 Mg; Procedure: Rehabilitation
- Placebo (Placebo Comparator): Week 2 after muscle strain injury Placebo pill, no active compounds 2x daily
  Interventions: Procedure: Rehabilitation; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen 500 Mg — Attenuating the sub-acute inflammatory processes to monitor potential beneficial tissue healing following a muscle strain injury
  Other Names: Anti-inflammatory Agents, Non-steroidal
  Arms: Anti-inflammatory medicine
Procedure: Rehabilitation — Rehabilitation after muscle strain injury
  Other Names: Physical therapy to stimulate tissue healing
Drug: Placebo — Sub-acute inflammatory processes not attenuated. Group will be treated as control to monitor tissue healing following a muscle strain injury without pharmacological intervention.
  Other Names: inert pills
  Arms: Placebo

SUMMARY:
Acute muscle strain injuries occur both during sports, in leisure time activities and during manual occupation and represent a major clinical challenge and has societal economic costs. The recovery time is long and a substantial injury recurrence is observed. Despite current best evidence rehabilitation with early mechanical loading, a significant loss of muscle mass, fatty infiltration and formation of scar tissue is reported.

Animal models and human in vitro experiments suggest that inflammation is vital in the early period after an injury, however an inhibition of inflammatory processes is beneficial for healing.

We investigate here whether a pharmacological inhibition of inflammatory pathways in the 2nd week following a muscle strain injury will provide a better clinical outcome and an advantageous cellular profile than rehabilitative training alone would.

DETAILED DESCRIPTION:
Injuries in skeletal muscle occur in sports, under recreational activities and during manual occupational work, and it represents both a significant clinical challenge and a burden for the individual in the form of long-term functional disability and pain, and for society causing a major economic cost (Ekstrand 2011). Traumatic muscle strain injuries occur most often in the hamstring and the calf region, are caused by high-force movements and most often result in a partial defect at the muscle-tendon (aponeurosis) interface (Tidball 1993, 2017). A major clinical challenge is that the recovery after a traumatic muscle strain injury is often long and in addition to this, substantial injury recurrence is observed. Several studies estimate that 80% of re-injuries occur at the site of the original injury (Wangensteen 2016).

It is known that early mechanical loading is important for shortening the period until pain-free return-to-sport (Bayer 2017). Whereas that study supports the role for mechanical loading in tissue repair and clinical recovery in the form of pain-free return to sports, early loading did not prevent muscle strength reduction and a significant loss of muscle mass in the injured muscle group, indicating that the recovery of the injured region is incomplete (Bayer 2018).

Experimental muscle injury precipitates an inflammatory response in the damaged tissue, which includes sequential infiltration of many cells and the release of inflammatory cytokines and growth factors (Chazaud 2016). Further, a study with human muscle cells and tissue after experimentally induced muscle injury found that a pro-inflammatory phase characterized by M1-macrophages was obligatory needed in the first 7 days after injury in order to initiate the healing process, manifested as proliferation capacity of the myogenic precursor cells (MPC) (Saclier 2013). It can be argued thus that a blockade of this proinflammatory phase would inhibit the healing process. In contrast, to advance the healing process after this initial pro-inflammatory phase, a switch to more anti-inflammatory activity - M2-macrophage activity - was needed in the later phase (7-14 days) to ensure differentiation of the MPC and thus a continued regeneration of tissue (Saclier2013). It is therefore possible that this anti-inflammatory stage is vital and that continued inflammation would cause an overall suboptimal healing response. Recently, a long-lasting inflammatory response after a muscle strain injury was reported. Based on analysis of injury exudates, very high levels of several pro-inflammatory factors were observed (Bayer 2019). Persistent presence of inflammation is linked to the development of fibrotic tissue changes in the long run (Wynn 2016) and importantly, fibrotic changes have been described following strain injuries (Bayer 2021, Silder 2008). Also, as prolonged elevated TNF-α (tumor necrosis factor-α) is known as an activator of the Nuclear Factor NF-κB pathway, this could cause stimulation of muscle atrophy related genes (Cohen 2015). It appears therefore clinically relevant to ensure that the pro-inflammatory phase following strain injuries is initially undisturbed, but the continuous pro-inflammatory phase is blunted to reduce the formation of fibrosis.

The aim of the present study is to test the hypothesis that an inhibition of inflammation, combined with the best standard training regimen in the later phase of recovery after injury (day 7-14) will provide a more optimal tissue recovery after injury than training alone will do.

The overall hypothesis is that administration of NSAID in the second week after an acute muscle strain injury in otherwise healthy humans, will be beneficial for tissue healing, characterized by an improved cellular composition allowing for less scar formation in the regeneration phase.

Participants will undergo a basic physical examination, including ultrasonographic scanning of the injured muscle site and fulfill questionnaire regarding previous injury history and present activities as well as symptoms.

Participants are then randomized to either placebo or NSAID treatment (Bonyl/ Naproxen 500 mg x 2 per day for 7 days) starting on day 7 and continued until day 14 post injury.

When participants are free of pain during movement including repeated explosive movements, the duration of the injury onset until full recovery is recorded (time to return to sports). Each participant will be followed by questionnaires for one year to record potential re-injuries.

Biopsies will be taken in week 1 post injury, before the pharmacological intervention, and in week 3 post injury, after the pharmacological intervention.

Biopsies will be analyzed by single nuclei RNA sequencing. Bioinformatics will be applied to investigate the distribution and number of cells in the injured muscle. Each biopsy will be compared to the control muscle (the same muscle as the injured one on the healthy, contralateral leg).

The biopsies will be obtained with a semi-automatic equipment that is routinely used to sample tendon tissue and tissue from chronic scar area in muscle (Bard Monopty) with a diameter of 1,6 mm a length of 10 mm.

ELIGIBILITY:
Inclusion Criteria:

* Sports-active individuals with an acute muscle train injury in either the hamstrings or calf muscle caused by an explosive movement (during sprinting, jumping etc)
* Age older than 18 years

Exclusion Criteria:

* Lack of hypoechoic/ hyperechoic area on ultrasound
* Diabetes type I and II
* Connective tissue disorders, rheumatism or any other chronic disease affecting the musculoskeletal system
* Anticoagulant medication
* Needle phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of anti-inflammatory medicine on cellular profile in skeletal muscle | 12 months
  Single-nuclei RNA sequencing (seq) of muscle tissue after a strain injury. Single nuclei RNA seq will be performed on biopsies obtained in week 1 after the strain injury. The cellular profile will be compared to the contralateral healthy muscle. Another biopsy, in both the injured and contralateral healthy muscle will be taken in week 3 post injury to investigate the effect of one week of Naproxen treatment versus inert placebo pills on the cellular profile measured with single nuclei RNA seq.

SECONDARY OUTCOMES:
Functional outcome performance | Up to 12 months
  Return-to-Sport. The time from onset of injury until the participants full and pain-free return to sport will be recorded.
Functional outcome re-injury rate | 12 months
  The number of re-injuries, participants sustain within 12 months after the initial strain injury will be recorded.
Functional outcome Patient Related Outcome Measures (PROM) | 12 months
  Participants will be asked to fill in a strain injury specific questionnaire as a "Patient related outcome measures ("PROM"). The questionnaire has 5 sub-categories including pain, symptoms, soreness, function during daily activities and sports and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Kjaer, DMSCi, Study Director — Bispebjerg Hospital

REFERENCES:
- [Background] Ekstrand J, Hagglund M, Walden M. Injury incidence and injury patterns in professional football: the UEFA injury study. Br J Sports Med. 2011 Jun;45(7):553-8. doi: 10.1136/bjsm.2009.060582. Epub 2009 Jun 23. PMID 19553225
- [Background] Wangensteen A, Tol JL, Witvrouw E, Van Linschoten R, Almusa E, Hamilton B, Bahr R. Hamstring Reinjuries Occur at the Same Location and Early After Return to Sport: A Descriptive Study of MRI-Confirmed Reinjuries. Am J Sports Med. 2016 Aug;44(8):2112-21. doi: 10.1177/0363546516646086. Epub 2016 May 16. PMID 27184543
- [Background] Chazaud B. Inflammation during skeletal muscle regeneration and tissue remodeling: application to exercise-induced muscle damage management. Immunol Cell Biol. 2016 Feb;94(2):140-5. doi: 10.1038/icb.2015.97. Epub 2015 Nov 3. PMID 26526620
- [Background] Saclier M, Yacoub-Youssef H, Mackey AL, Arnold L, Ardjoune H, Magnan M, Sailhan F, Chelly J, Pavlath GK, Mounier R, Kjaer M, Chazaud B. Differentially activated macrophages orchestrate myogenic precursor cell fate during human skeletal muscle regeneration. Stem Cells. 2013 Feb;31(2):384-96. doi: 10.1002/stem.1288. PMID 23169615
- [Background] Wynn TA, Vannella KM. Macrophages in Tissue Repair, Regeneration, and Fibrosis. Immunity. 2016 Mar 15;44(3):450-462. doi: 10.1016/j.immuni.2016.02.015. PMID 26982353
- [Background] Bayer ML, Hoegberget-Kalisz M, Svensson RB, Hjortshoej MH, Olesen JL, Nybing JD, Boesen M, Magnusson SP, Kjaer M. Chronic Sequelae After Muscle Strain Injuries: Influence of Heavy Resistance Training on Functional and Structural Characteristics in a Randomized Controlled Trial. Am J Sports Med. 2021 Aug;49(10):2783-2794. doi: 10.1177/03635465211026623. Epub 2021 Jul 15. PMID 34264782
- [Background] Bayer ML, Magnusson SP, Kjaer M; Tendon Research Group Bispebjerg. Early versus Delayed Rehabilitation after Acute Muscle Injury. N Engl J Med. 2017 Sep 28;377(13):1300-1301. doi: 10.1056/NEJMc1708134. No abstract available. PMID 28953439
- [Background] Bayer ML, Hoegberget-Kalisz M, Jensen MH, Olesen JL, Svensson RB, Couppe C, Boesen M, Nybing JD, Kurt EY, Magnusson SP, Kjaer M. Role of tissue perfusion, muscle strength recovery, and pain in rehabilitation after acute muscle strain injury: A randomized controlled trial comparing early and delayed rehabilitation. Scand J Med Sci Sports. 2018 Dec;28(12):2579-2591. doi: 10.1111/sms.13269. Epub 2018 Aug 16. PMID 30043997
- [Background] Silder A, Sherry MA, Sanfilippo J, Tuite MJ, Hetzel SJ, Heiderscheit BC. Clinical and morphological changes following 2 rehabilitation programs for acute hamstring strain injuries: a randomized clinical trial. J Orthop Sports Phys Ther. 2013 May;43(5):284-99. doi: 10.2519/jospt.2013.4452. Epub 2013 Mar 13. PMID 23485730
- [Background] Cohen S, Nathan JA, Goldberg AL. Muscle wasting in disease: molecular mechanisms and promising therapies. Nat Rev Drug Discov. 2015 Jan;14(1):58-74. doi: 10.1038/nrd4467. PMID 25549588
- [Background] Bayer ML, Bang L, Hoegberget-Kalisz M, Svensson RB, Olesen JL, Karlsson MM, Schjerling P, Hellsten Y, Hoier B, Magnusson SP, Kjaer M. Muscle-strain injury exudate favors acute tissue healing and prolonged connective tissue formation in humans. FASEB J. 2019 Sep;33(9):10369-10382. doi: 10.1096/fj.201900542R. Epub 2019 Jun 18. PMID 31211922